CLINICAL TRIAL: NCT02270515
Title: Bringing Care to Patients: A Patient-Centered Medical Home for Kidney Disease
Brief Title: Bringing Care to Patients: Patient-Centered Medical Home for Kidney Disease
Acronym: PCMH-KD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Denise M. Hynes, PhD, MPH, RN, Professor, College of Medicine; Research Affiliate, School of Public Health; and, Biomedical Informatics Core Director, Center for Clinical and Translational Sciences (CCTS),, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IH-12-11-5420
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: ESRD
Keywords: Patient-Centered Care; Medical Home
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PCMH-KD dialysis care (Experimental): Dialysis care team is expanded to include a primary care doctor, nurse coordinator, community health worker, and pharmacist. Enrolled patients are observed for an initial baseline period receiving care under the usual dialysis care model called the 'usual dialysis care phase'.
  Interventions: Other: Patient-Centered Medical Home for Kidney Disease (PCMH-KD)

INTERVENTIONS:
Other: Patient-Centered Medical Home for Kidney Disease (PCMH-KD) — A PCMH-KD enhances the usual dialysis care team by adding a primary care doctor, pharmacist, nurse coordinator and community health worker to the care team.

SUMMARY:
This study will implement and evaluate a patient-centered medical home for kidney disease (PCMH-KD) compared to the usual model of dialysis care. Patients will be observed for an initial baseline period under the usual care model and then the usual dialysis care team will be expanded to include a pharmacist, community health worker, nurse coordinator and a primary care doctor. Outcomes of interest will be assessed at baseline and then every 6 months after the PCMH-KD intervention commences.

DETAILED DESCRIPTION:
Patients with end-stage renal disease (ESRD), have unique and complex care needs associated with renal disease and common comorbidities (e.g., diabetes, hypertension), and under the current care model, receive fragmented care from multiple providers at multiple locations. ESRD patients typically spend three to five hours undergoing dialysis three days a week. Scheduling and traveling to other appointments are difficult to manage, increase patient and caregiver burden, and reduce patients' quality of life. These challenges keep many ESRD patients from receiving care for other conditions outside of the dialysis setting, resulting in higher rates of complications, and emergent healthcare use.

The patient-centered medical home (PCMH) model has been proposed as a solution to patients with complex needs such as those with ESRD. The purpose of this project is to compare a PCMH model of care with the usual care of ESRD patients and their caregivers. We propose to enhance the usual care team for ESRD patients by providing a primary care doctor in the context of regularly scheduled dialysis sessions and by adding community health workers to help support patients and their caregivers. Patient and family stakeholders and care team members will assist in the design and refinement of the PCMH model.

We plan to implement this model at the University of Illinois Hospital and Health Sciences System (UIHS) dialysis center and a local Fresenius Medical Care dialysis center. Patients receiving dialysis at participating centers will receive an initial comprehensive care visit followed by ongoing care from a multispecialty provider team during the patients' regularly scheduled dialysis visits. Each patient's care team will include a kidney doctor, a primary care doctor, a nurse coordinator, a dialysis nurse, a dietician, a pharmacist, a social worker, and a community health worker. The primary care doctor will be available in the dialysis clinic to provide general and preventive care to the patient before or after dialysis sessions. This doctor would also coordinate care with other specialists/clinicians on the patient's care team. The trained, bilingual (English/Spanish) community health worker will assist with making and rescheduling appointments, obtaining transportation, and reinforcing education components.

We expect that this approach will increase patient access to care for other conditions and will increase care coordination and communication among members of the patient's care team. These improvements could potentially increase the likelihood of preventing complications or identifying problems earlier and allow for a more successful treatment. We expect that this enhanced care team will reduce emergency room visits and hospitalizations for dialysis patients. In addition, we anticipate that the addition of community health workers to the clinical team will help support and educate patients and their caregivers and as a result, patient quality of life will improve and caregiver burden may be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Current patient receiving hemodialysis at two participating dialysis centers who are able to provide informed consent

Exclusion Criteria:

* Not a patient at one of the two participating dialysis centers or not able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2013-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Hynes, PhD, MPH, RN, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - Fresenius Medical Care Chicago Westside dialysis center, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System dialysis center, Chicago, Illinois

REFERENCES:
- [Background] Porter AC, Fitzgibbon ML, Fischer MJ, Gallardo R, Berbaum ML, Lash JP, Castillo S, Schiffer L, Sharp LK, Tulley J, Arruda JA, Hynes DM. Rationale and design of a patient-centered medical home intervention for patients with end-stage renal disease on hemodialysis. Contemp Clin Trials. 2015 May;42:1-8. doi: 10.1016/j.cct.2015.02.006. Epub 2015 Feb 28. PMID 25735489
- [Background] Cukor D, Cohen LM, Cope EL, Ghahramani N, Hedayati SS, Hynes DM, Shah VO, Tentori F, Unruh M, Bobelu J, Cohen S, Dember LM, Faber T, Fischer MJ, Gallardo R, Germain MJ, Ghahate D, Grote N, Hartwell L, Heagerty P, Kimmel PL, Kutner N, Lawson S, Marr L, Nelson RG, Porter AC, Sandy P, Struminger BB, Subramanian L, Weisbord S, Young B, Mehrotra R. Patient and Other Stakeholder Engagement in Patient-Centered Outcomes Research Institute Funded Studies of Patients with Kidney Diseases. Clin J Am Soc Nephrol. 2016 Sep 7;11(9):1703-1712. doi: 10.2215/CJN.09780915. Epub 2016 May 19. PMID 27197911
- [Background] Hynes DM, Buscemi J, Quintiliani LM; Society of Behavioral Medicine Health Policy Committee. Society of Behavioral Medicine (SBM) position statement: SBM supports increased efforts to integrate community health workers into the patient-centered medical home. Transl Behav Med. 2015 Dec;5(4):483-5. doi: 10.1007/s13142-015-0340-1. Epub 2015 Aug 28. PMID 26622920
- [Result] Hynes DM, Fischer MJ, Schiffer LA, Gallardo R, Chukwudozie IB, Porter A, Berbaum M, Earheart J, Fitzgibbon ML. Evaluating a novel health system intervention for chronic kidney disease care using the RE-AIM framework: Insights after two years. Contemp Clin Trials. 2017 Jan;52:20-26. doi: 10.1016/j.cct.2016.10.003. Epub 2016 Oct 18. PMID 27769897

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The PCMH-KD model was implemented at two dialysis centers, an academic dialysis center and a private dialysis center. Patients were recruited, screened and enrolled at both sites. After consenting, study participants completed a baseline survey and on a rolling basis three follow-up interviews at six, twelve, and eighteen months.
Pre-assignment Details: Clinical data (six months prior to enrollment date) was collected from the electronic medical record for all participants to compare the "usual care" for enrolled patients with the care received during the PCMH-KD intervention.
Groups:
- PCMH-KD Dialysis Care: Dialysis care team is expanded to include a primary care doctor, nurse coordinator, community health worker, and a pharmacist.
  Patient-Centered Medical Home for Kidney Disease (PCMH-KD): A PCMH-KD enhances the usual dialysis care team by adding a primary care doctor, pharmacist, nurse coordinator and community health worker to the care team.
Period: Intervention Period 1: 0-6 Months
Arm/Group | PCMH-KD Dialysis Care
Started | 175
Completed | 159
Not Completed | 16
Not completed — Withdrawal by Subject | 1
Not completed — No longer patient at study site | 5
Not completed — Received transplant | 3
Not completed — Death | 7
Period: Intervention Period 2: 6-12 Months
Arm/Group | PCMH-KD Dialysis Care
Started | 159
Completed | 127
Not Completed | 32
Not completed — Withdrawal by Subject | 2
Not completed — No longer patient at study site | 7
Not completed — Received transplant | 1
Not completed — Death | 5
Not completed — Intervention ended before follow-up | 17
Period: Intervention Period 3: 12-18 Months
Arm/Group | PCMH-KD Dialysis Care
Started | 127
Completed | 103
Not Completed | 24
Not completed — Withdrawal by Subject | 1
Not completed — No longer patient at study site | 2
Not completed — Received transplant | 2
Not completed — Death | 3
Not completed — Intervention ended before follow-up | 16

BASELINE CHARACTERISTICS:
Groups:
- PCMH-KD Dialysis Care: Enrolled patients had access to an expanded care team inlcuding a primary care doctor, nurse coordinator, community health worker, and pharmacist.
Arm/Group | PCMH-KD Dialysis Care
Number analyzed (Participants) | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Hispanic/other category consist of Hispanic and participants of unidentified race
  Participants
    Race/Ethnicity: African-American | 86
    Race/Ethnicity: Hispanic/other | 89
Region of Enrollment [Number; unit: participants]
  United States | 175
Interview language [Count of Participants; unit: Participants]
  English | 117
  Spanish | 58
Race/ethnicity*language [Count of Participants; unit: Participants]
  African-American | 86
  Hispanic/other, English interview | 31
  Hispanic, Spanish interview | 58
Primary language [Count of Participants; unit: Participants]
  English | 107
  Spanish/other | 54
  Both equally | 14
Marital status [Count of Participants; unit: Participants]
  Single, never married | 70
  Married/Living with a partner | 62
  Widowed | 22
  Separated, divorced | 21
Children under 18 yr in household [Count of Participants; unit: Participants]
  No children under 18 yr in household | 132
  1 child under 18 yr in household | 22
  ≥ 2 children under 18 yr in household | 21
Education [Count of Participants; unit: Participants]
  Not HS graduate | 62
  HS graduate/GED | 100
  Bachelor's degree | 13
Employment [Count of Participants; unit: Participants] — Population: No Response: 1 participant
  Participants
    number analyzed (Participants) | 174
    Full-time/Self-employed | 16
    Part-time | 15
    Not employed | 143
Income [Count of Participants; unit: Participants]
  Less than $20,000 | 108
  $20,000-$39,999 | 30
  ≥ $40,000 | 22
  Refused | 15
Dialysis History [Mean (Standard Deviation); unit: years] — Population: Missing dialysis information for one (1) study participant.
  years
    Years on dialysis: number analyzed (Participants) | 174
    Years on dialysis | 4.4 (5.2)
    Years at current center: number analyzed (Participants) | 174
    Years at current center | 3.3 (4.4)
Primary transportation to clinic [Count of Participants; unit: Participants]
  Car (drive or ride) | 87
  Transit (L train or bus) | 14
  Medicar (Medicaid) | 42
  PACE paratransit/door to door | 17
  Other | 15
Insurance (any type) [Count of Participants; unit: Participants]
  Yes | 158
  No | 17
Comorbidities [Count of Participants; unit: Participants]
  None | 15
  1 | 55
  2 to 3 | 91
  4 to 7 | 14
Stressful life events (e.g. hospitalization, loss of employment or family member) in past 6 months [Count of Participants; unit: Participants]
  Yes | 79
  No | 96
Regular doctor (Primary Care Physician) [Count of Participants; unit: Participants]
  Has regular personal doctor | 104
  No regular personal doctor | 71
Primary Care Assessment Survey (PCAS) [Mean (Standard Deviation); unit: units on a scale] — Primary Care Assessment Survey (PCAS) assesses patient satisfaction for five (5) primary care characteristics Longitudinal Continuity, Comprehensive Knowledge, Communication, Interpersonal Treatment, and Integration of Care. PCAS scale scores ranges from 0 to 100. Higher scores are more positive (better outcome). Population: 1. Longitudinal Continuity, Comprehensive Knowledge, Communication and Interpersonal Treatment scores are calculated for patients who reported having a regular personal doctor.
  2. Integration of Care is calculated for patients who reported having a regular personal doctor and reported receiving referrals.
  3. Numbers differ due to missing data.
  units on a scale
    Longitudinal Continuity: number analyzed (Participants) | 104
    Longitudinal Continuity | 52.9 (37.2)
    Comprehensive Knowledge: number analyzed (Participants) | 104
    Comprehensive Knowledge | 65.4 (21.3)
    Communication: number analyzed (Participants) | 104
    Communication | 74.3 (18.8)
    Interpersonal Treatment: number analyzed (Participants) | 104
    Interpersonal Treatment | 75.2 (17.3)
    Integration of Care: number analyzed (Participants) | 64
    Integration of Care | 67.8 (22.2)
Self-Efficacy for Managing Chronic Disease (SEMCD) [Mean (Standard Deviation); unit: units on scale] — This 6-item scale measures confidence in common activities needed to managechronic conditions. Scores range from 1 to 10. Higher scores indicate higher self-efficacy. Population: Missing data for (1) study participant.
  units on scale
    number analyzed (Participants) | 174
    (all) | 7.2 (2.0)
Chronic Hemodialysis Knowledge Survey (CHeKS) [Mean (Standard Deviation); unit: units on scale] — Chronic Hemodialysis Knowledge Survey (CHeKS) measures patient's hemodialysis knowledge. Score ranges from 0 to 100. Mean score closer to 100 means better outcome/score. Population: Missing data for one (1) study participant.
  units on scale
    number analyzed (Participants) | 174
    (all) | 51.8 (15.7)
Health Literacy [Count of Participants; unit: Participants] — Health literacy score ranges from 3 to 15 with lower score meaning higher health literacy.
  Participants
    Adequate (3-8) | 106
    Inadequate/marginal (9-15) | 69

OUTCOME MEASURES:

1. Primary Outcome: Kidney Disease Quality of Life (KDQOL-36) Mean Scale Scores at Baseline, 6, 12 and 18 Months: Unadjusted
Description: Quality of life (QOL) was measured using the Kidney Disease Quality of Life-36 (KDQOL-36) survey, a kidney-disease-specific quality of life instrument that assesses five domains: general physical health, mental health, disease burden, disease symptoms, and disease effects. For all KDQOL scales, a higher score indicates better quality of life. All domain scales can range from 0-100.
Time Frame: Baseline (0) to 18 months
Population: Overall number of participants analyzed are the number who completed the KDQOL at each visit. They differ slightly from the number of participants in the flow chart due to missing KDQOL data. Ns are slightly lower for some scale scores due to missing items (see below).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline: KDQOL collected at Baseline
- 6 Months: KDQOL collected at 6 months
- 12 Months: KDQOL collected at 12 months
- 18 Months: KDQOL collected at 18 months
Arm/Group | Baseline | 6 Months | 12 Months | 18 Months
Number analyzed (Participants) | 174 | 153 | 125 | 103
units on a scale
  Physical Component Summary (PCS): number analyzed (Participants) | 172 | 152 | 125 | 102
  Physical Component Summary (PCS) | 35.5 (10.2) | 38.4 (11.4) | 36.3 (11.2) | 36.8 (11.2)
  Mental Component Summary (MCS): number analyzed (Participants) | 172 | 152 | 125 | 102
  Mental Component Summary (MCS) | 49.2 (10.6) | 50.4 (11.3) | 51.8 (10.2) | 52.4 (9.7)
  Burden of Kidney Disease | 46.5 (27.1) | 48.8 (26.7) | 49.6 (23.3) | 51.2 (30.3)
  Symptoms/Problems of Kidney Disease | 76.5 (15.9) | 79.9 (14.2) | 79.7 (13.6) | 76.8 (16.7)
  Effects of Kidney Disease | 72.3 (20.6) | 76.3 (20.6) | 78.3 (18.9) | 76.1 (20.1)

2. Primary Outcome: Kidney Disease Quality of Life (KDQOL-36) Mean Scale Scores at Baseline, 6, 12 and 18 Months: Adjusted
Description: Quality of life (QOL) was measured using the Kidney Disease Quality of Life-36 (KDQOL-36) survey, a kidney-disease-specific quality of life instrument that assesses five domains: general physical health, mental health, disease burden, disease symptoms, and disease effects. For all KDQOL scales, a higher score indicates better quality of life. All domain scales can range from 0-100.
  Adjusted means are from random-intercept linear mixed models with an AR(1) covariance pattern in the residual, adjusted for baseline age, sex, race (AA, all other), interview language, dialysis vintage (months), site, education (not HS grad, HS grad), marital status (married or living with partner, other), self-reported diabetes at baseline, PCP at baseline, urea reduction ratio (URR), hemoglobin (g/dL), and albumin (g/dL). The 3 lab values are time-varying covariates.
Time Frame: Baseline (0) to 18 months
Population: Ns shown in the table are the number of records at each visit with data for the KDQOL scale score and all covariates. All available records were used to estimate the adjusted means. For all scales, N=173 participants; 2 were excluded due to missing data for covariates: dialysis vintage and PCP at baseline.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | 6 Months | 12 Months | 18 Months
Number analyzed (Participants) | 172 | 147 | 125 | 102
units on a scale
  Physical Component Summary (PCS): number analyzed (Participants) | 170 | 146 | 125 | 101
  Physical Component Summary (PCS) | 35.7 (0.9) | 38.3 (1.0) | 36.0 (1.0) | 36.7 (1.1)
  Mental Component Summary (MCS): number analyzed (Participants) | 170 | 146 | 125 | 101
  Mental Component Summary (MCS) | 48.9 (0.9) | 50.1 (1.0) | 51.4 (1.0) | 51.7 (1.1)
  Burden of Kidney Disease | 45.8 (2.4) | 48.4 (2.5) | 49.0 (2.5) | 49.7 (2.7)
  Symptoms/Problems of Kidney Disease | 77.1 (1.3) | 79.6 (1.4) | 79.3 (1.5) | 76.4 (1.5)
  Effects of Kidney Disease | 73.0 (1.8) | 77.2 (1.9) | 79.6 (2.0) | 76.9 (2.1)

3. Primary Outcome: Estimated KDQOL-36 Scale Score Change for Each 6-month Period and 0-18 Months: Adjusted Random-intercept Models
Description: as for outcome 1
Time Frame: Baseline (0) to 18 months
Population: All records with data for the KDQOL scale score (dependent variable) and covariates were included in the analysis. Two participants were excluded due to missing data for covariates: dialysis vintage and PCP at baseline. The previous table (adjusted means) shows the number of records with complete data for each visit.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Change 0-6 Months: Change of mean score from Baseline (0) to 6 months
- Change 6-12 Months: Change of mean score from 6 months to 12 months
- Change 12-18 Months: Change of mean score from 12 months to 18 months
- Change 0-18 Months: Change of mean score from Baseline (0) to 18 months
Arm/Group | Change 0-6 Months | Change 6-12 Months | Change 12-18 Months | Change 0-18 Months
Number analyzed (Participants) | 173 | 173 | 173 | 173
units on a scale
  Physical Component Summary (PCS) | 2.6 (0.8) | -2.3 (0.9) | 0.7 (1.0) | 1.0 (1.0)
  Mental Component Summary (MCS) | 1.2 (1.0) | 1.3 (1.0) | 0.3 (1.1) | 2.8 (1.1)
  Burden of Kidney Disease | 2.6 (2.0) | 0.6 (2.0) | 0.6 (2.2) | 3.8 (2.1)
  Symptoms/Problems of Kidney Disease | 2.6 (1.1) | -0.4 (1.2) | -2.9 (1.3) | -0.7 (1.3)
  Effects of Kidney Disease | 4.3 (1.5) | 2.4 (1.6) | -2.8 (1.8) | 3.9 (1.7)
Statistical Analysis 1: Comparison: Change 0-6 Months; PCS: From random-intercept linear mixed models with an AR(1) covariance pattern in the residual, adjusted for baseline age, sex, race (AA, all other), interview language, dialysis vintage (months), site, education (not HS grad, HS grad), marital status (married or living with partner, other), self-reported diabetes at baseline, PCP at baseline, urea reduction ratio (URR), hemoglobin (g/dL), and albumin (g/dL). The 3 lab values are time-varying covariates; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — This is the PCS KDQOL Subscale p-value for change in 0-6 months shown in Primary Outcome table 3
Statistical Analysis 2: Comparison: Change 0-6 Months; MCS: From random-intercept linear mixed models with an AR(1) covariance pattern in the residual, adjusted for baseline age, sex, race (AA, all other), interview language, dialysis vintage (months), site, education (not HS grad, HS grad), marital status (married or living with partner, other), self-reported diabetes at baseline, PCP at baseline, urea reduction ratio (URR), hemoglobin (g/dL), and albumin (g/dL). The 3 lab values are time-varying covariates; Test type: Superiority or Other; p = 0.23, Mixed Models Analysis — This is the MCS KDQOL Subscale p-value for change in 0-6 months shown in Primary Outcome table 3
Statistical Analysis 3: Comparison: Change 0-6 Months; Burden: From random-intercept linear mixed models with an AR(1) covariance pattern in the residual, adjusted for baseline age, sex, race (AA, all other), interview language, dialysis vintage (months), site, education (not HS grad, HS grad), marital status (married or living with partner, other), self-reported diabetes at baseline, PCP at baseline, urea reduction ratio (URR), hemoglobin (g/dL), and albumin (g/dL). The 3 lab values are time-varying covariates; Test type: Superiority or Other; p = 0.18, Mixed Models Analysis — This is the Burden KDQOL Subscale p-value for change in 0-6 months shown in Primary Outcome table 3
Statistical Analysis 4: Comparison: Change 0-6 Months; Symptoms: From random-intercept linear mixed models with an AR(1) covariance pattern in the residual, adjusted for baseline age, sex, race (AA, all other), interview language, dialysis vintage (months), site, education (not HS grad, HS grad), marital status (married or living with partner, other), self-reported diabetes at baseline, PCP at baseline, urea reduction ratio (URR), hemoglobin (g/dL), and albumin (g/dL). The 3 lab values are time-varying covariates; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis — This is the Symptoms KDQOL Subscale p-value for change in 0-6 months shown in Primary Outcome table 3
Statistical Analysis 5: Comparison: Change 0-6 Months; Effects: From random-intercept linear mixed models with an AR(1) covariance pattern in the residual, adjusted for baseline age, sex, race (AA, all other), interview language, dialysis vintage (months), site, education (not HS grad, HS grad), marital status (married or living with partner, other), self-reported diabetes at baseline, PCP at baseline, urea reduction ratio (URR), hemoglobin (g/dL), and albumin (g/dL). The 3 lab values are time-varying covariates; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — This is the Effects KDQOL Subscale p-value for change in 0-6 months shown in Primary Outcome table 3
Statistical Analysis 6: Comparison: Change 6-12 Months; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis — This is the PCS KDQOL Subscale p-value for change in 6-12 months shown in Primary Outcome table 3
Statistical Analysis 7: Comparison: Change 6-12 Months; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.21, Mixed Models Analysis — This is the MCS KDQOL Subscale p-value for change in 6-12 months shown in Primary Outcome table 3
Statistical Analysis 8: Comparison: Change 6-12 Months; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.77, Mixed Models Analysis — This is the Burden KDQOL Subscale p-value for change in 6-12 months shown in Primary Outcome table 3
Statistical Analysis 9: Comparison: Change 6-12 Months; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.77, Mixed Models Analysis — This is the Symptoms KDQOL Subscale p-value for change in 6-12 months shown in Primary Outcome table 3
Statistical Analysis 10: Comparison: Change 6-12 Months; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.14, Mixed Models Analysis — This is the Effects KDQOL Subscale p-value for change in 6-12 months shown in Primary Outcome table 3
Statistical Analysis 11: Comparison: Change 12-18 Months; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.45, Mixed Models Analysis — This is the PCS KDQOL Subscale p-value for change in 12-18 months shown in Primary Outcome table 3
Statistical Analysis 12: Comparison: Change 12-18 Months; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.79, Mixed Models Analysis — This is the MCS KDQOL Subscale p-value for change in 12-18 months shown in Primary Outcome table 3
Statistical Analysis 13: Comparison: Change 12-18 Months; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.77, Mixed Models Analysis — This is the Burden KDQOL Subscale p-value for change in 12-18 months shown in Primary Outcome table 3
Statistical Analysis 14: Comparison: Change 12-18 Months; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis — This is the Symptoms KDQOL Subscale p-value for change in 12-18 months shown in Primary Outcome table 3
Statistical Analysis 15: Comparison: Change 12-18 Months; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.12, Mixed Models Analysis — This is the Effects KDQOL Subscale p-value for change in 12-18 months shown in Primary Outcome table 3
Statistical Analysis 16: Comparison: Change 0-18 Months; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.29, Mixed Models Analysis — This is the PCS KDQOL Subscale p-value for change in 0-18 months shown in Primary Outcome table 3
Statistical Analysis 17: Comparison: Change 0-18 Months; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis — This is the MCS KDQOL Subscale p-value for change in 0-18 months shown in Primary Outcome table 3
Statistical Analysis 18: Comparison: Change 0-18 Months; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.08, Mixed Models Analysis — This is the Burden KDQOL Subscale p-value for change in 0-18 months shown in Primary Outcome table 3
Statistical Analysis 19: Comparison: Change 0-18 Months; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.61, Mixed Models Analysis — This is the Symptoms KDQOL Subscale p-value for change in 0-18 months shown in Primary Outcome table 3
Statistical Analysis 20: Comparison: Change 0-18 Months; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis — This is the Effects KDQOL Subscale p-value for change in 0-18 months shown in Primary Outcome table 3

ADVERSE EVENTS:
Time Frame: Baseline to 18 months
Groups:
- PCMH-KD Dialysis Care: Dialysis care team is expanded to include a primary care doctor, nurse coordinator, community health worker, and pharmacist.
  Patient-Centered Medical Home for Kidney Disease (PCMH-KD): A PCMH-KD enhances the usual dialysis care team by adding a primary care doctor, pharmacist, nurse coordinator and community health worker to the care team.
Arm/Group | PCMH-KD Dialysis Care
Serious Adverse Events (participants affected / at risk) | 0/175
Other Adverse Events (participants affected / at risk) | 0/175

LIMITATIONS AND CAVEATS:
Subjects were not randomized to the intervention, although their experience prior to the intervention (baseline measures) served as the historical control. Only two sites were included in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No